CLINICAL TRIAL: NCT06005584
Title: Spinal Cord Stimulation to Reduce Imbalance and Falls in Parkinson's Disease
Brief Title: Spinal Cord Stimulation for Gait Dysfunction in Parkinson's Disease
Acronym: SCORE-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 22CX7894
Record Dates: First submitted 2023-01-27; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Spinal Cord Stimulation; Parkinson's; Gait Disorders
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- High Frequency SCS (Active Comparator): Participants will be randomly assigned to this arm for up to 6 weeks
  Interventions: Device: Spinal Cord Stimulation - High Frequency SCS
- Burst SCS (Active Comparator): Participants will be randomly assigned to this arm for up to 6 weeks
  Interventions: Device: Spinal Cord Stimulation - Burst SCS
- Sham SCS (Sham Comparator): Participants will be randomly assigned to this arm for up to 6 weeks
  Interventions: Device: Spinal Cord Stimulation - Sham SCS

INTERVENTIONS:
Device: Spinal Cord Stimulation - High Frequency SCS — High Frequency-SCS consists of delivering electrical stimulation at frequencies equal to or greater than 1kHz.
  This intervention will last up to 6 weeks.
  Arms: High Frequency SCS
Device: Spinal Cord Stimulation - Burst SCS — Burst SCS consists of closely spaced, high frequency stimuli delivered to the spinal cord.
  This intervention will last up to 6 weeks.
  Arms: Burst SCS
Device: Spinal Cord Stimulation - Sham SCS — This intervention will last up to 6 weeks.
  Arms: Sham SCS

SUMMARY:
Parkinson's disease (PD) is the second commonest neurodegenerative disorder, affecting over 145,000 people in the UK. Initially, PD patients experience slowness of movements, limb stiffness, and tremor.

With progressive loss of neurons over time, many patients start to experience balance and walking problems, and falls, which are resistant to currently available treatments. Falls can lead to fractures and nursing home admission, and can significantly shorten patients' life expectancy.

In this pilot study, the investigators will investigate the effects of spinal cord stimulation (SCS) on gait and balance in PD. Some open-labelled studies have shown possible beneficial effects of SCS in PD, although it is uncertain which type of PD patients will benefit most and which stimulation parameters work best. The investigators will assess the effects of SCS on posture and gait using a series of clinical, laboratory, imaging, and wearable measurements.

The participants will receive a percutaneous implantation of a spinal cord stimulator to minimise the possible adverse effects related to the surgery.

The SCS will start one month after surgery. The investigators will use a double-blind cross-over design. The participants will receive three different stimulation parameters, including sham stimulation, in a randomised order. The participants and the assessors will be blinded to the stimulation parameters.

DETAILED DESCRIPTION:
The investigators aim to recruit up to 8 people with Parkinson's with significant gait dysfunction which is resistant to medical therapy to this study. All participants will receive implantation of a spinal cord stimulator at T8-10 levels. The procedure will be done percutaneously. The spinal cord stimulation will be commenced 2-4 weeks after surgery to allow time for recovery.

Participants will receive 3 different stimulation parameters in randomised order as outlined below:

1. Burst stimulation
2. High frequency stimulation
3. Sham stimulation Each parameter will last for up to 6 weeks. Both the patients and the researchers assessing the patients will be blinded to the settings parameters. At baseline and at the end of each stimulation settings, the participants will undergo a series of assessments (see secondary outcomes). At the end of the cross-over blinded period, the participants will be unblinded and offered to continue with the parameter that offered most symptomatic relief. The participants will then continue in this setting in an open label phase for another 10 weeks before their final assessment at 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45 ≤ X ≤ 85
* PD diagnosis based on UK Parkinson's disease society brain bank criteria
* Significant gait dysfunction, particularly freezing of gait, which is resistant to optimal medical therapy
* Hoen and Yahr stage: 2-4 (in ON state)
* Stable dopaminergic treatment for at least two weeks before enrolment.
* Can provide informed consent

Exclusion Criteria:

* Atypical or secondary parkinsonism e.g. vascular, drug-induced
* Major focal brain disorders (including malignancy or stroke)
* Recent (within 3 months)/current use of acetylcholinesterase inhibitors or antidopaminergic drugs
* Concomitant treatment with deep brain stimulation
* Neurological, vestibular, visual or orthopaedic diagnosis significantly interfering with gait
* Pregnant women or planning to become pregnant
* Significant chronic back pain
* Spinal anatomical abnormalities precluding SCS surgery
* Major cognitive or psychiatric illness
* Concomitant or recent (less than 4 months) enrolment in an interventional research trial.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Incidence of Treatment-Emergent Adverse Events | Day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Safety of a 28-week SCS Intervention will be assessed by measuring the number of participants with adverse events that are related to treatment
Number of Participants with Incidence of Serious Adverse Events | Day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Safety of a 28-week SCS Intervention will be assessed by measuring the number of participants with serious adverse events
Number of Participants that complete the study | Day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Safety of a 28-week SCS Intervention will be assessed by measuring the number of participants that complete the study

SECONDARY OUTCOMES:
1. Mean change from baseline to week 28 in participant scores on the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part 3 motor subsection in the "OFF" and "ON" medication state | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Motor symptoms will be measured using the MDS-UPDRS part 3 motor subsection. Part III of the scale will be completed at baseline, visit 1 (1 day post-surgery), visit 2 (6 weeks post-surgery), visit 3 (12 weeks post-surgery), visit 4 (18 weeks post-surgery), visit 4 (28 weeks post-surgery).
  The scale consists of four parts; Part I "Non-motor experiences of daily living" (13 questions), Part II "Motor Experiences of daily living" (13), Part III "Motor Examination" (33) and Part IV "Motor Complications" (6).
  Each question has five responses that are linked to common clinical terms: 0=Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. "Slight" refers to symptoms with sufficiently low frequency/intensity to cause no impact on function; "Mild" refers to symptoms of frequency/intensity sufficient to cause modest impact on function; "Moderate" refers to symptoms sufficiently frequent/intense to impact considerably, but not prevent, function; "Severe" refers to symptoms that prevent function.
Change in Hoehn and Yahr Scoring Scale | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Scores range: 1-5. Higher scores mean a worse outcome.
Change in New Freezing of Gait Questionnaire | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  The new freezing of gait questionnaire is a measure of freezing severity (total score range: 0-28) wherein higher scores represent worse freezing behaviour.
  The outcome measures represent the change in freezing of gait questionnaire score from pre-intervention (baseline visit) to each post-intervention time point. A larger, positive value represents a greater reduction in freezing severity and a better outcome.
Changes in 10 meter walk test (10MW) performance (sec) | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Change in the duration to walk 10 meters (in seconds), both in ON-medication. A longer duration to perform the task represents a more impaired mobility.
Changes in Timed Up and Go (TUG) test Performance (sec) | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Change in the duration to perform the Timed-Up and Go (TUG) test in seconds, with and without a cognitive dual task, in ON-medication. The Timed Up and Go performance is a measure of mobility, and a longer duration to perform the task represents a more impaired mobility.
Changes in 360° turning performance (sec) | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Change in the duration to turn 360° in place in ON medication, with and without a cognitive dual task. A longer duration to perform the task represents a more impaired mobility.
Mean change in objective, unsupervised quantification of participant motor impairment, using motion sensors | Baseline, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Motor impairment will be determined based on recordings using five sensors (both arms and legs, and lower back) for the entire duration of the trial (PD Monitor, PD Neuroelectrics). Sensors will be placed before the SCS surgery and after each change in SCS parameter, up to the end of the open label phase (28 weeks).
Change in balance: objective measure of sway velocity on a force platform (metre/sec) | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Sway will be measured on a force platform before and after each SCS parameter change, up to 28 weeks post-intervention. Sway metric (sway velocity) will be collected at each time point in five different conditions, namely while standing on an hard surface with eyes open (condition 1) and closed (condition 2), on a soft surface with eyes open (condition 3) and closed (condition 4), and while tandem standing with eyes open (condition 5).
Changes in Non-motor Symptoms of PD | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Non Motor Symptoms Scale (NMSS) Minimum: 0, maximum: 360, higher score values indicate a worse outcome.
Changes in Quality of Life Measured by a 39-item Parkinson's Disease Questionnaire (PDQ-39) | Baseline, day 1 post-surgery, week 6 post-surgery, week 12 post-surgery, week 18 post-surgery, week 28 post-surgery
  Parkinson's Disease Questionnaire - 39 (PDQ-39) is a self-administered questionnaire. It comprises of 39 questions, relating to eight key areas of health and daily activities, including both Motor and Non-motor symptoms. It is scored on a scale of zero to 100, with lower scores indicating better health and high scores more severe symptoms in change from Baseline to end of Maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Yen Tai, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Group data can be made available upon request, following completion and publication of results